CLINICAL TRIAL: NCT01167166
Title: A Phase 1/2, Single Arm Study To Assess the Efficacy and Safety of Rigosertib (ON 01910.Na) Administered as 72-Hour and 120-Hour Continuous Intravenous Infusions Every Other Week for Two Cycles Then as Twice Daily Oral Capsules Given Continuously in Patients With Relapsed/Refractory Acute Myeloid or Lymphocytic Leukemia or Transformed Myeloproliferative Neoplasms
Brief Title: Safety and Efficacy of 72-hour and 120-hour Infusion of Rigosertib in Acute Myeloid Leukemia (AML) and Acute Lymphoid Leukemia (ALL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-19
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Acute Myelocytic Leukemia; Acute Lymphocytic Leukemia; Myeloproliferative Disease; Chronic Myeloid Leukemia
Keywords: Acute Myelocytic Leukemia; Acute Lymphocytic Leukemia; Myeloproliferative Disease; Myelofibrosis; Essential thrombocythemia; Polycythemia vera; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rigosertib (Experimental): Patients will receive 2400 mg dose of rigosertib as a intravenous continuous infusion over 24 hours for 72 to 120 consecutive hours every 2 weeks for the first 4 weeks then will receive oral rigosertib at a 560 mg twice-daily dose as capsules taken continuously.
  Interventions: Drug: rigosertib

INTERVENTIONS:
Drug: rigosertib — The dose of rigosertib will be 2400 mg/24h as an intravenous continuous infusion over 72 or 120 hours every 2 weeks for 2 cycles then as oral capsules administered at a dose of 560 mg twice daily on a continuous basis.
  Other Names: rigosertib sodium

SUMMARY:
For patients with leukemia who have not responded to or have progressed after an initial response to standard therapy, therapeutic options are limited. Although responses to standard regimens do occur, durable remissions are achieved infrequently and current regimens are not curative in the majority of patients. Identification of active agents in patients with relapsed Acute Myeloid Leukemia (AML) ultimately affords the potential for use upfront as a component of induction regimens that may translate to improved outcome. Therefore, development of new agents is of critical importance. This study will look at a new, investigational agent, ON 01910.Na, to determine if it has the potential to help Patients with AML and Acute Lymphocytic Leukemia (ALL) and transformed Myeloproliferative Neoplasms.

DETAILED DESCRIPTION:
This is a single center, open-label, phase 1/2 study in which 2 to 34 patients with refractory acute myeloid or lymphocytic leukemia or transformed myeloproliferative neoplasms (MPNs)who meet all other inclusion/exclusion criteria will be administered a daily dose of 2400 mg ON 01910.Na dose as a intravenous continuous infusion (IVCI) over 24 hours for 72 to 120 consecutive hours every 2 weeks for the first 4 weeks then will receive oral rigosertib at a 560 mg twice-daily dose as capsules taken continuously.

In the phase 1 component of the trial, a standard dose escalation scheme will be followed with the enrolment of at least three patients treated with a daily dose of 2400 mg ON 01910.Na IVCI over 24 hours for 72 hours. The dose escalation scheme will follow a traditional dose escalation rule, also known as the "3+3" rule:

If none of the initial three patients treated in the 72-hour cohort experience dose-limiting toxicity (DLT), during the first two 2-week cycles, then a new cohort of three patients will be treated at the same 2400 mg/24h daily dose but for an increased 120 hours duration.

DLT is defined as an adverse event possibly related to ON 01910.Na that is:

* Grade ≥ 3 non-hematological toxicity other than nausea, vomiting, diarrhea, fever, esophagitis/dysphagia
* Grade ≥ 3 nausea and vomiting uncontrolled by antiemetics; grade ≥ 3 diarrhea uncontrolled by antidiarrheal agents; grade ≥ 3 drug-induced fever uncontrolled by antipyretics; grade ≥3 metabolic abnormalities that are not controlled by optimal supportive care measures
* Grade ≥ 3 stomatitis and/or esophagitis/dysphagia lasting > 3 days
* Marrow cellularity <5% on day 42 or later (6 weeks) from start of therapy without evidence of leukemia

If one of the three patients in the 72-hour cohort experiences a DLT during the first two cycles, then three additional patients will be treated for the same 72 hours duration. Escalation to the 120-hour cohort will proceed only if no more than one of the six patients treated in the 72-hour cohort experiences a DLT.

If two or more patients in the 72-hour cohort experience DLT during the first two cycles, then the maximum tolerated dose (MTD) will have been exceeded, no further dosing extension will occur, and a full safety review will determine if further enrollment of patients will proceed.

If none of the initial three patients in the 120-hour cohort experiences DLT during the first two cycles, this regimen will be confirmed as the Maximum Tolerated Dose (MTD) and no further dose escalation will occur.

If one of the three patients in the 120-hour cohort experiences DLT during the first two cycles, then three additional patients will be treated for the same duration. If no more than one patient experiences a DLT, the 120-hour regimen will be confirmed as the Maximum Tolerated Dose (MTD) and no further dose escalation will occur.

If two or more patients in the 120 hours cohort experience DLT during the first two cycles, then the maximum tolerated dose (MTD) will be determined to be 2400 mg/24h administered for 72 hours every other week.

Once the phase 1 portion of the study is completed, accrual to the phase 2 portion will begin. Patients treated at the MTD during the phase 1 portion will be included in the phase 2 component and will be evaluated for response and secondary end points.

The total study duration is 30 weeks, which includes a 2-week screening phase, a 24-week dosing phase (4-week rigosertib CIV administration, followed by 20 weeks of oral rigosertib administration), and a 4-week follow-up phase that begins after the last dose of rigosertib. Beginning at week 5, patients will be assessed for response every time a complete blood count (CBC) is performed and followed up.

Patients who achieve by week 24 a response or stabilization of their disease are eligible to receive an additional 24 weeks of rigosertib at the same dose and will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented or cytologically confirmed diagnosis of one of the following hematological malignancies:

   * Acute myelocytic leukemia (AML) refractory to standard induction treatment, or relapsed after standard therapy (including transformed myeloproliferative diseases with at least 10% blasts in bone marrow and chronic myeloid leukemia in a blast phase)
   * Transformed myeloproliferative neoplasms (MPNs; i.e., myelofibrosis, essential thrombocythemia (ET), polycythemia vera (PV)) with at least 10% blasts in bone marrow and chronic myeloid leukemia in a blast phase refractory or relapsing after standard therapy
   * Acute lymphocytic leukemia (ALL) refractory to induction treatment, or relapsed after standard therapy
2. Patients should not have received any prior chemotherapy for their leukemia or transformed MPN within 14 days and should have recovered from any toxicity related to prior chemotherapy to at least grade 1. In the presence of rapidly proliferating disease, patients can be included after a washout period of 7 days. Hydroxyurea can be administered as clinically indicated, and no washout is required.
3. Patients may not be candidates for, or must have declined, bone marrow transplantation from an HLA-identical donor in the immediate future (ie, within 4 weeks) or other chemotherapeutic regimens known to produce consistent remissions.
4. Patients with known meningeal infiltration may be enrolled only if radiation has been completed, and a clearing of peripheral blood blasts has been noted. Intrathecal therapy can be continued if judged to be in the best interest of the patient to prevent recurrence, provided there is no toxicity associated with it and there has been clearance of blasts in the cerebrospinal fluid.
5. ECOG Performance Status 0, 1 or 2.
6. Willing to adhere to the prohibitions and restrictions specified in this protocol.
7. Patient must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
2. Known HIV-1 seropositivity.
3. Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
4. Uncontrolled active systemic infection not adequately responding to appropriate therapy.
5. Total bilirubin ≥ 1.5 mg/dL not related to hemolysis or Gilbert's disease.
6. ALT or AST ≥ 2.5 X ULN.
7. Serum creatinine ≥ 2.0 mg/dL.
8. Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 Meq/L).
9. Female patients who are pregnant or lactating; Male patients with female sexual partners who are unwilling to follow the strict contraception requirements (condom use). Patients of reproductive potential who do not agree to use adequate contraceptive before entry and throughout the study; Female patients with reproductive potential who do not have a negative serum or urine beta-HCG pregnancy test at screening.
10. Major surgery without full recovery or major surgery within 3 weeks of rigosertib treatment start.
11. Uncontrolled hypertension (defined as a systolic pressure equal to or greater than 160 and/or a diastolic pressure equal to or greater than 100).
12. New onset seizures (within 3 months prior to the first dose of rigosertib) or poorly controlled seizures
13. Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy.
14. Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 8 months
  DLT: adverse event possibly related that is:
  * Grade ≥ 3 non-hematological toxicity other than nausea, vomiting, diarrhea, fever, esophagitis/dysphagia
  * Grade ≥ 3 nausea and vomiting uncontrolled by antiemetics; grade ≥ 3 diarrhea uncontrolled by antidiarrheal agents; grade ≥ 3 drug-induced fever uncontrolled by antipyretics; grade ≥3 metabolic abnormalities that are not controlled by optimal supportive care measures
  * Grade ≥ 3 stomatitis and/or esophagitis/dysphagia lasting > 3 days
  * Marrow cellularity <5% on day 42 or later (6 weeks) from start of therapy without evidence of leukemia
Change in bone marrow blast cell and peripheral blood counts at 5, 13 and 25 weeks | 18 months
  Determine the clinical response rate (complete or partial remission) according to response criteria in patients with relapsed/refractory acute myeloid or lymphocytic leukemia (1 Cheson BD, Bennett JM, Kopecky KJ, et al. Revised Recommendations of the International Working Group for Diagnosis, Standardization or Response Criteria, Treatment Outcomes and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. JCO 21:4642, 2003).

SECONDARY OUTCOMES:
Concentration of ON 01910.Na in plasma | Week 1 and Week 3
  Blood samples to determine concentration of rigosertib in plasma will be collected at 6 hours after the start of the second 24-hour infusion (Day 2) at Weeks 1 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Patient and cancer information on M. D. Anderson Cancer Center web site. — http://www.mdanderson.org/patient-and-cancer-information/index.html